CLINICAL TRIAL: NCT03850613
Title: Alleviating Caregivers' Stress Through an E-painting Mobile Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Angela Leung, Associate Professor, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: G-YBWL
Record Dates: First submitted 2018-12-19; First posted 2019-02-22 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Caregivers; Anxiety
Keywords: caregivers, stress, anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The recruited subjects (n=30) will be assigned to the intervention group and use the newly developed app for 8 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Participants in the intervention arm download the E-painting mobile app and use this app to make their own painting.
  Interventions: Behavioral: E-painting mobile app

INTERVENTIONS:
Behavioral: E-painting mobile app — The subjects can use the newly developed mobile app to draw their own pictures at the time convenient to them.

SUMMARY:
This study aims to develop a mobile app for caregivers and tests its feasibility for a period of 8 weeks. A mixed-method study design with both qualitative and quantitative components will be used. A maximum of 36 caregivers will be involved in the six focus groups. Each focus group interview will involve 6 caregivers of persons with dementia. Another 30 caregivers will be involved in the 8-week trial use of the app. Each focus group interview will last for about 1.5 hours, facilitated by a moderator. Before and after the 8-week trial use of the app, four outcome measures (Zarit Burden Interview, Self-rated Health, Patient Health Questionnaire, and Modified Medical Outcome Study Social Support Survey) will be taken. This study will provide evidence of the feasibility of the use of the newly developed app among caregivers.

DETAILED DESCRIPTION:
Background Caregivers of persons with dementia experience tremendous stress Caregivers of persons with dementia (PWD) in Hong Kong reported high level of stress due to caregiving (Cheung et al., 2015). Caregiver stress was defined as "an unequal distribution of responsibilities on the caregiver as a result of caring for someone with a prolonged impairment" (Pearlin et al., 1990 cited in Llanque et al., 2016). Providing care to PWD persons imposed tremendous stress on caregivers as PWD often performed problematic behaviours that might affect others (Kang et al., 2006). PWD's dependency in activities of daily living, severity and frequency of behavioural symptoms was found to be significantly associated with caregivers' depressive symptoms (Lee et al., 2017). Another source of stress was caregivers' feeling of overload, which was considered as subjective stressor (Son et al., 2007).

Use of mobile applications in stress management Mobile applications (apps) have been developed in stress management. Persons suffered from post-traumatic stress disorders have been selected as targeted population to assess feasibility and acceptability of apps to manage acute stress or stress symptoms (Kuhn et al., 2014). From the users' perspective (as stated in focus group interviews), using app was considered as 'acceptable and helpful' tool for stress management (Kuhn et al., 2014). Activities could be scheduled by the app and this arrangement was welcome by app users (Kuhn et al., 2014). Apps are considered as potentially effective self-management tool for persons suffered from stress (Kuhn et al., 2014).

New feature of the mobile app: e-painting Evidence had shown that intervention of art therapy reduced stress symptoms among paediatric patients (Chapman et al., 2001), working adults (Karpaviciute & Macijauskiene, 2016), and older adults (Walker et al., 2016). Group interactions among participants in art therapy contributed to its effectiveness, thus group therapy was recommended as 'best practice' (Spiegel et al., 2006). Painting (or visual art production) is recommended because looking at painting (or cognitively evaluated artwork) does not show similar effect on stress reduction in adulthood (Bolwerk et al., 2014). Using functional MRI (fMRI), Bolwerk and team (2014) found that those who participated in visual art production showed greater spatial improvement in functional connectivity of posterior cingulated cortex to the frontal and parietal cortices after the intervention than those who cognitively evaluated artwork at a museum. This implied that painting, but not viewing art work, had effect on psychological resilience in adulthood (Bolwerk and team, 2014). A review (Slayton et al., 2010) summarised that a brief period of painting significantly reduced anxiety score (Sandmire et al., 2012; Curry & Kasser, 2005), distress (Franks & Whitaker, 2007), depression (Gussak, 2006) but increased mental alertness and sociability (Rusted, Sheppard, & Waller, 2006).

Based on the knowledge in the production of painting and its possible impacts on caregivers' emotion (anxiety, stress, depression) and sociability, we plan to develop a mobile application which allows caregivers to create their own e-paintings and share with others.

Objectives of the study

1. To identify caregivers' preferred functions of the app and training needed to use the app;
2. To assess the trial process and procedures (estimate the recruitment rate, dropout rate, the compliance of emotional assessments in the app);
3. To collect app users' comments on the use of the app after the 8-week trial;
4. To examine the consistency of the effects of the app intervention on emotion.

Methods This study adopts a mixed method (qualitative and quantitative method).

Qualitative component comprises of six focus group (FG) interviews. FG 1-3 aim to explore the caregivers' preferences of the features of the e-painting mobile app. FG 4-6 aim to collect the app users' views on the use of the app after the trial period of 8 weeks.

Guiding questions for Focus Group 1-3:

1. What functions are preferred by the caregivers in the e-painting app?
2. What kind of training do caregivers need before they use the e-painting app?
3. What kind of follow-up do caregivers expect after using this app? Analytical results of their paintings in form of a prop-up message? Connection to health professionals who could provide help to the caregivers?

Guiding questions for Focus Group 4-6:

1. What did the app users (caregivers) think about this app?
2. What did the app users like or dislike most about the app?
3. What feature should be added to the app so as to support the app users?
4. Did the app users enjoy the use of this app to draw their paintings? Why?

Quantitative component of the study is the trial run of the app over a period of 8 weeks with 30 caregivers. Participants will be asked to download the app to their mobile phone and use the app at least two times per week. They will be asked to go through a set of emotion assessments in the app before and after the 8-week trial. The following measures will be included in the emotional assessments:

1. Caregivers' level of stress (measured by a 11-item Zarit Burden Interview, CZBI-Short, Tang et al., 2015) (Primary outcome)
2. Self-rated health status (measured by the 1-item self-rated health likert scale) (Secondary outcome)
3. Depressive symptoms (measured by a 9-item Patient Health Questionnaire (PHQ-9, Cheng & Cheng, 2007) (Secondary outcome)
4. Instrumental and emotional social support (measured by a 8-item Modified Medical Outcome Study Social Support Survey (mMOS-SS, Moser et al., 2012) (Secondary outcome)

E-paintings will be analysed by a certified art therapist through discussions with the participants. Data about colour hue, saturation and brightness will be analysed. Data will be collected in recruitment rate of caregivers who are willing to join the study, the dropout rate at the end of the 8-week trial, and the compliance rate of emotional assessments in the app. Frequency of the participation in e-painting will be collected. Comparison of the app users' stress level, depressive level, self-rated health status and social support before and after the trial will be made.

Subjects. A maximum of 36 caregivers will be involved in the six focus groups. Each focus group interview will involve 6 caregivers of persons with dementia. Another 30 caregivers will be involved in the 8-week trial of the app.

Expected deliverables

1. A e-painting mobile app for caregiver to reduce stress;
2. A presentation in an international conference (reporting app users' comments on the use of the app after the 8-week trial);
3. A paper in an international peer-refereed journal (reporting caregivers' preferred functions of the app, the training needed to use the app, the recruitment rate of caregivers to the study, the dropout rate of participation in the 8-week trial, the compliance of emotional assessments in the app and the consistency of the effects of the app intervention on emotion).

ELIGIBILITY:
Inclusion criteria:

* aged 18 or above
* provide direct care to a person with dementia
* able to read and communicate in Chinese

Exclusion criteria:

* have fever or influenza symptoms at the time of recruitment
* being hospitalized
* living in a residential care home

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Caregivers' level of stress | right after the 8-week intervention
  this will be measured by a 11-item Zarit Burden Interview (CZBI-Short) (Tang et al., 2015)

SECONDARY OUTCOMES:
Self-rated health status | right after the 8-week intervention
  This will be measured by the 1-item self-rated health likert scale
Depressive symptoms | right after the 8-week intervention
  This will be measured by a 9-item Patient Health Questionnaire (PHQ-9) (Cheng & Cheng, 2007)
Instrumental and emotional social support | right after the 8-week intervention
  This will be measured by a 8-item Modified Medical Outcome Study Social Support Survey (mMOS-SS) (Moser et al., 2012)

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Llanque S, Savage L, Rosenburg N, Caserta M. Concept Analysis: Alzheimer's Caregiver Stress. Nurs Forum. 2016 Jan-Mar;51(1):21-31. doi: 10.1111/nuf.12090. Epub 2014 May 1. PMID 24787468
- [Result] Bolwerk A, Mack-Andrick J, Lang FR, Dorfler A, Maihofner C. How art changes your brain: differential effects of visual art production and cognitive art evaluation on functional brain connectivity. PLoS One. 2014 Jul 1;9(7):e101035. doi: 10.1371/journal.pone.0101035. eCollection 2014. PMID 24983951
- [Result] Cheung KS, Lau BH, Wong PW, Leung AY, Lou VW, Chan GM, Schulz R. Multicomponent intervention on enhancing dementia caregiver well-being and reducing behavioral problems among Hong Kong Chinese: a translational study based on REACH II. Int J Geriatr Psychiatry. 2015 May;30(5):460-9. doi: 10.1002/gps.4160. Epub 2014 Jul 12. PMID 25043378
- [Result] Karpaviciute S, Macijauskiene J. The Impact of Arts Activity on Nursing Staff Well-Being: An Intervention in the Workplace. Int J Environ Res Public Health. 2016 Apr 19;13(4):435. doi: 10.3390/ijerph13040435. PMID 27104550
- [Result] Kuhn E, Greene C, Hoffman J, Nguyen T, Wald L, Schmidt J, Ramsey KM, Ruzek J. Preliminary evaluation of PTSD Coach, a smartphone app for post-traumatic stress symptoms. Mil Med. 2014 Jan;179(1):12-8. doi: 10.7205/MILMED-D-13-00271. PMID 24402979
- [Result] Lee J, Sohn BK, Lee H, Seong S, Park S, Lee JY. Impact of Behavioral Symptoms in Dementia Patients on Depression in Daughter and Daughter-in-Law Caregivers. J Womens Health (Larchmt). 2017 Jan;26(1):36-43. doi: 10.1089/jwh.2016.5831. Epub 2016 Aug 9. PMID 27505267
- [Result] Son J, Erno A, Shea DG, Femia EE, Zarit SH, Stephens MA. The caregiver stress process and health outcomes. J Aging Health. 2007 Dec;19(6):871-87. doi: 10.1177/0898264307308568. PMID 18165286